CLINICAL TRIAL: NCT05087979
Title: Use of Stable Airway Management Device in Monitored Anesthesia Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HM20022338
Record Dates: First submitted 2021-10-08; First posted 2021-10-21 (Actual); Results first posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia
Keywords: monitored anesthesia care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Intervention (Experimental): An investigational device will be used to hold patient's head and airway in a stable position.
  Interventions: Device: Stable airway management (SAM) device
- Standard of care (No Intervention): Pillows and towels will be used to hold patient's head and airway in a stable position.

INTERVENTIONS:
Device: Stable airway management (SAM) device — SAM is positioning device that will maintain patient's head, neck, and therefore their airway in the correct position during their procedure.
  Arms: Intervention

SUMMARY:
The aim of this study is to determine if the Stable Airway Management device (SAM) is safe in maintaining the airway in a stable, non-obstructing position during anesthetic cases requiring monitored anesthesia care (MAC).

DETAILED DESCRIPTION:
Patients undergoing monitored anesthesia care as part of a procedure will be invited to participate in the study.

The stable airway management (SAM) device is an investigational device used to hold patient's head and airway in a stable position during a MAC procedure. An investigational device means it has not been approved by the U. S. Food and Drug Administration (FDA). In this study, the SAM will be compared to the standard of anesthesia care which consists of supporting patient's head, neck, and shoulders with pillows and towels when placing them in the correct position for the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing MAC anesthesia in the supine position
2. Patients able to give informed consent

Exclusion Criteria:

1. Age < 18 years
2. Less than 88% oxygen saturation on room air
3. Non-elective procedures
4. Case duration > 180 minutes
5. Presence of a cervical spine injury, instability, or cervical spine collar
6. Patients with airway, facial, or other anatomy deemed inappropriate for SAM use by anesthesiologist
7. General anesthesia as primary anesthetic
8. Prisoners
9. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Visnal Yajnik, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Standard of Care
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0
Not completed — Converted to general anesthesia | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Standard of Care | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Median (Full Range); unit: years] | 61 [26 to 78] | 61 [38 to 84] | 61 [26 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 7 | 9 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Total Apneic Events /Total Number Requiring Airway Manipulation
Description: total number of apneic events greater than 20 seconds per 15-minute intervals, requiring airway manipulation - The median value of airway manipulations will be reported for each arm, along with the range of manipulations (low-high) for each study arm will be reported.
Time Frame: Up to 6 hours
Measure: Median (Full Range); unit: Number of airway manipulations
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 19 | 20
Number of airway manipulations | 2 [0 to 10] | 1 [0 to 11]

2. Primary Outcome: Number of Subjects Converted From MAC to General Anesthesia
Description: Number of participants converted from MAC to general anesthesia for airway-related complications
Time Frame: Up to 6 hours
Measure: Number; unit: participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 19 | 20
participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 3-4 days post procedure
Description: Post-procedure safety monitoring: patient self report. Patients rated their level of discomfort in the jaw, neck, and head from the start of the procedure up until day 3 of post-procedure
Arm/Group | Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-11-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT05087979/Prot_000.pdf